CLINICAL TRIAL: NCT03982459
Title: Acceptability and Effectiveness of a Novel Internet -Based Decision-Support Aid Based on the NCCN Non-Small Cell Lung Cancer Patient Guidelines
Brief Title: National Comprehensive Cancer Network (NCCN) Decision Support Tool for Patients With NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14655
Record Dates: First submitted 2019-05-27; First posted 2019-06-11 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision support tool (Experimental): Participants receive training in use of a decision support tool by a trained coordinator.
  Interventions: Behavioral: Decision support tool

INTERVENTIONS:
Behavioral: Decision support tool — Internet-Based, interactive decision support tool

SUMMARY:
This study involves the evaluation of a decision support tool, based on the patient version of the NCCN guidelines, for the non-small cell lung cancer patient population.

DETAILED DESCRIPTION:
This study involves the evaluation of a decision support tool, based on the patient version of the NCCN guidelines, for the non-small cell lung cancer patient population. The decision support tool is offered by a trained coordinator to the patient and then utilized during an initial consultation. Patients complete forms before and after the visit indicating their level of decisional conflict, satisfaction, and satisfaction with decision. Pre-determined indices of quality of care were also collected by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Over age of 18
* Able to provide informed consent
* Able to use a web-based interface
* Histologically proven or clinically apparent diagnosis of non-small cell lung cancer
* Newly diagnosed, with new primary occurrence of NSCLC, or diagnosed with a new recurrence or new progression of existing disease, and not yet treated for the new problem
* Being seen in consultation at thoracic oncology clinics

Exclusion Criteria:

* Unable to fill out questionnaires
* Already treated for the current diagnosis of a new primary occurrence of NSCLC, or already treated for the new recurrence or new progression of existing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request.
Access Criteria: Requests for datasets should be sent to the Principal Investigator for review and approval for dissemination.

REFERENCES:
- [Background] Wu SY, Lazar AA, Gubens MA, Blakely CM, Gottschalk AR, Jablons DM, Jahan TM, Wang VEH, Dunbar TL, Wong ML, Chan JW, Guthrie W, Belkora J, Yom SS. Evaluation of a National Comprehensive Cancer Network Guidelines-Based Decision Support Tool in Patients With Non-Small Cell Lung Cancer: A Nonrandomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e209750. doi: 10.1001/jamanetworkopen.2020.9750. PMID 32997124

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision Support Tool: Participants receive training in use of a decision support tool by a trained coordinator at a single clinic visit.
Period: Overall Study
Arm/Group | Decision Support Tool
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 42
Age, Continuous [Mean (Full Range); unit: years] | 68 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 51
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Quality of Care on Selected National Comprehensive Cancer Center (NCCN) Recommendations
Description: Participants explored individually tailored decision trees derived from the NCCN guidelines. Six benchmarks of quality care derived from the guidelines were evaluated: (1) documented smoking cessation counseling in active smokers, (2) adjuvant chemotherapy for patients with stage IB to IIB NSCLC after surgery, (3) pathologic mediastinal staging in patients with stage III NSCLC before surgery, (4) pathologic mediastinal staging in patients with stage III NSCLC before nonsurgical management, (5) definitive chemoradiotherapy for patients with stage III NSCLC not undergoing surgery, and (6) molecular testing for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) alterations for patients with stage IV NSCLC. Because the decision trees were tailored, not all participants evaluated all 6 benchmarks. The percentage of participants who interacted with each benchmark and demonstrated quality of care will be reported.
Time Frame: 1 Day
Population: Nine participants were missing survey results preventing calculation for this measure
Measure: Number; unit: percentage of participants
Groups:
- Decision Support Tool: Patients in this single-arm study all receive training in use of a decision support tool by a trained coordinator.
  decision support tool: computerized online decision support tool
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 65
percentage of participants
  Documented smoking cessation counseling or intervention in active smokers: number analyzed (Participants) | 5
  Documented smoking cessation counseling or intervention in active smokers | 80
  Adjuvant chemotherapy for participants with stage IB-IIB disease following surgery: number analyzed (Participants) | 7
  Adjuvant chemotherapy for participants with stage IB-IIB disease following surgery | 0
  Pathologic mediastinal staging completed before surgery for patients with stage III disease: number analyzed (Participants) | 2
  Pathologic mediastinal staging completed before surgery for patients with stage III disease | 50
  Pathologic mediastinal staging before treatment initiation for stage III not undergoing surgery: number analyzed (Participants) | 14
  Pathologic mediastinal staging before treatment initiation for stage III not undergoing surgery | 28.6
  Initial chemoradiotherapy for participants with stage III disease not undergoing surgery: number analyzed (Participants) | 14
  Initial chemoradiotherapy for participants with stage III disease not undergoing surgery | 64.3
  Testing for EGFR or ALK gene alteration status for participants with stage IV disease: number analyzed (Participants) | 23
  Testing for EGFR or ALK gene alteration status for participants with stage IV disease | 91.3

2. Secondary Outcome: Median Change in Decisional Conflict Scale (DCS) Score Over Time
Description: Change in level of decisional conflict will be assessed by the DCS completed before and after consultation. The DCS is a scale designed to measure participants' uncertainty in making health-related decisions, factors contributing to uncertainty, and participants perceived effective decision-support. The DCS has a total of 16 items and uses a five-point Likert scale for each item. The total score ranging from 0-64 is divided by 16 and then multiplied by 25 to calculate a final total score with 0 indicating low conflict and 100 indicating high conflict. The median change in score over time and the interquartile range will be reported.
Time Frame: 1 Day
Population: Nine participants did not complete the questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 65
score on a scale | 20 [3 to 34]

3. Secondary Outcome: Median Scores by Item on the Satisfaction With Health Care Decision Questionnaire
Description: The Patient Satisfaction with Health Care Decision (SWD) Questionnaire is a six-item survey with item responses ranging from 1 -5 with a higher value indicating a higher degree of satisfaction or agreement with the statement.
  The median score of each item and the interquartile range will be reported.
Time Frame: 1 Day
Population: Six participants did not complete the questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 70
score on a scale
  I am satisfied that I am adequately informed about the issues important to my decision | 4 [4 to 5]
  The decision I made was the best decision possible for me personally | 4 [3 to 5]
  I am satisfied that my decision was consistent with my personal values | 4 [3 to 5]
  I expect to successfully carry out (or continue to carry out) the decision I made | 4 [4 to 5]
  I am satisfied that this was my decision to make | 4 [4 to 5]
  I am satisfied with my decision | 4 [4 to 5]

4. Secondary Outcome: Number of Participants by Response on the Decisional Support Preference Questionnaire (DMPQ)
Description: Participants preferred style of decision making with their physician will be assessed using the Decision Making Preference Questionnaire (DMPQ). The DMPQ consists of a single question with five choices, ranging from a preference to have the doctor make all of the decisions (passive) to the patient making all of the decisions themselves about their treatment (active) or a combination of shared decision making ranging from the most passive in self-decision making preference to the most active in self-decision making. The number of participants by response will be reported.
Time Frame: 1 Day
Population: Five participants did not complete the questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 71
Participants
  Doctor should make the decisions | 5
  Doctor should make the decisions but strongly consider my opinion | 12
  Doctor and I should make the decisions together | 39
  I should make decisions but strongly consider the doctor's opinion | 13
  I should make the decision | 2

5. Secondary Outcome: Median Total Score on the Quality of Life by the Functional Assessment of Cancer Therapy-Lung (FACT-L) Questionnaire
Description: The Functional Assessment of Cancer Therapy-Lung (FACT-L) Scale is a 36-item self-report instrument that measures multidimensional quality of life for patients with lung cancer. Each item is rated on a 5-point Likert scale ranging from 0 = "Not at all" to 4 = "Very much" with a total score range of 0-144, and higher scores indicating a better quality of life.
Time Frame: 1 Day
Population: Two participants did not complete the questionnaire.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 74
score on a scale | 67 [61 to 75]

6. Secondary Outcome: Median Scores on the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy Lung Symptom Index (NFLSI-17)
Description: The NCCN/FACT Lung Cancer Symptom Index-17 (NFLSI-17) is a brief symptom index for patients with advanced lung cancer. The NFLSI-17 is a 17-item patient-reported questionnaire. Each item is rated on a 5-point Likert scale ranging from 0 = "Not at all" to 4 = "Very much" with a total score range of 0-68. The questionnaire includes three subscales: Disease-Related Subscale, Treatment Side Effects, and Functional Well-Being with higher scores indicating lower overall symptoms.
Time Frame: 1 Day
Population: data not collected
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants With Reported Agreement at Post Consultation With Physician
Description: The percentage of participants who completed the post-consultation questionnaire and reported achieving agreement on treatment recommendations between the participants and the physician with respect to treatments discussed and recommended, prognosis, and expected tolerance will be reported.
Time Frame: 1 Day
Population: Only 45 participants completed the questionnaire
Measure: Number; unit: percentage of participants
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 45
percentage of participants | 93.3

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Decision Support Tool
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03982459/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03982459/ICF_001.pdf